CLINICAL TRIAL: NCT04408521
Title: Effect of Long-lasting EEG-Neurofeedback on Attention Control and Impulsivity in Adult Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Effects of a Novel Neurofeedback Protocol on ADHD Subcomponents
Acronym: NFB@HOME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Nader Perroud, MD, Associate Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-01029; SNCTP000002260 (Registry Identifier: Kofam.ch (Koordinationsstelle Forschung am Menschen))
Record Dates: First submitted 2020-05-12; First posted 2020-05-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Electroencephalography; Alpha Rhythm; Attention; Impulsive Behavior; Neurofeedback
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEUROFEEDBACK (Experimental): Participants undergo individual at home sessions of 45-minute video-replay of popular TV series while recording their 1-channel EEG using a portable system. Self-regulation of alpha rhythm is reflected in the dynamically varying opacity of the video replay window, i.e. the window would turn lighter/darker and reveal/obscure video content during episodes of low/high alpha amplitude, respectively.
  Interventions: Other: NEUROFEEDBACK
- CONTROL (Placebo Comparator): Participants undergo individual at home sessions of 45-minute video-replay of popular TV series while recording their 1-channel EEG using a portable system. The recording is passive without real-time EEG neurofeedback (i.e. constant brightness and volume).
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: NEUROFEEDBACK — EEG recording during alpha-related TV viewing
  Arms: NEUROFEEDBACK
Other: CONTROL — EEG recording during passive TV viewing
  Arms: CONTROL

SUMMARY:
Mounting evidence suggests that closed-loop brain-training, commonly known as neurofeedback (NFB), may represent a new therapeutic opportunity for patients with Attentional Deficit/Hyperactivity Disorder (ADHD), which manifests as difficulties with attention and inhibitory control. In this context, the investigators have focused on an attention-enhancing form of NFB based on the EEG alpha rhythm, known to influence sensory detection and attention. In light of recent evidence showing that both attention and impulsivity can be modified with a single-session of alpha-NFB, the objective is to determine whether these effects stabilize in the long-term, after multiple, daily sessions of training at home.

A short- (single-session) and a long-term (multi-session) experimental design will be used to collect EEG, behavioral, and clinical data pre-to-post NFB. The single-blind study will recruit 48 adult ADHD participants randomly assigned to either NEUROFEEDBACK or CONTROL groups. Each participant will undergo individual at home sessions of 45-minute video-replay of popular television (TV) series while recording their 1-channel EEG (30 sessions, 5 sessions/week, 6 weeks total). In the NEUROFEEDBACK group, self-regulation of alpha rhythm will be reflected in the dynamically varying opacity of the video-replay window, i.e. the window would turn lighter/darker and reveal/obscure video content during episodes of low/high alpha amplitude, respectively. In the CONTROL group, the recording will be passive without real-time EEG neurofeedback (i.e. constant brightness and volume). Before and after at home training, each participant will have two visits in the lab: (1) complete clinical and neuropsychological evaluation and (2) EEG session including resting state and task-related EEG before and after a short NFB intervention (30 minutes). For the CONTROL group participants, the latter will be replaced by a sham intervention utilizing non-contingent feedback.

Given that stronger alpha rhythmicity is associated with increases in inhibitory/excitatory balance, it is expected that alpha-NFB (i) will homeostatically normalize alpha rhythm power and (ii) the degree of normalization will be a dimensional predictor of individual improvement in behavioral and clinical measures of executive function, impulsivity and inattention. These results should lay the foundation for building neurocognitive treatments, by harnessing neuroplasticity mechanisms intrinsic to the brain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD
* Currently stabilized (euthymic)
* General good health
* Normal or corrected-to normal visual acuity

Exclusion Criteria:

* Mood Disorders
* PTSD
* Borderline Personality Disorder
* Substance Use Disorder
* Structural Brain Abnormalities
* Cerebrovascular Disease
* Epilepsy
* Stroke
* Head Trauma
* Cardiovascular Disease
* Renal Failure
* Hepatic Dysfunction
* Impaired visual acuity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in assessor-evaluated clinical ADHD status | Change between day 10 pre-intervention and day 10 post-intervention
  Change in adult ADHD Child Evaluation (ACE+) scoring (min = 0, max = 36, higher score = worse outcome)
Change in self-reported clinical ADHD status | Change between day 10 pre-intervention and day 10 post-intervention
  Change in adult ADHD Self-Report Scale (ASRS) scoring (min = 0, max = 72, higher score = worse outcome)
Change in Alpha Spectral Power | Change between day 2 pre-intervention and day 2 post-intervention
  Absolute and relative spectral alpha power in the 8-12 Hz frequency range at rest (microvolts)
Change in reaction time at the Continuous Performance Task (CPT) | Change between day 2 pre-intervention and day 2 post-intervention
  Reaction time and reaction time variability (milliseconds)
Change in error rates at the CPT | Change between day 2 pre-intervention and day 2 post-intervention
  Number of omission and commission errors

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dayer, MD, PhD, Study Director — University of Geneva & University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arns M, de Ridder S, Strehl U, Breteler M, Coenen A. Efficacy of neurofeedback treatment in ADHD: the effects on inattention, impulsivity and hyperactivity: a meta-analysis. Clin EEG Neurosci. 2009 Jul;40(3):180-9. doi: 10.1177/155005940904000311. PMID 19715181
- [Background] Ergenoglu T, Demiralp T, Bayraktaroglu Z, Ergen M, Beydagi H, Uresin Y. Alpha rhythm of the EEG modulates visual detection performance in humans. Brain Res Cogn Brain Res. 2004 Aug;20(3):376-83. doi: 10.1016/j.cogbrainres.2004.03.009. PMID 15268915
- [Background] Macdonald JS, Mathan S, Yeung N. Trial-by-Trial Variations in Subjective Attentional State are Reflected in Ongoing Prestimulus EEG Alpha Oscillations. Front Psychol. 2011 May 10;2:82. doi: 10.3389/fpsyg.2011.00082. eCollection 2011. PMID 21687452
- [Background] Micoulaud-Franchi JA, Geoffroy PA, Fond G, Lopez R, Bioulac S, Philip P. EEG neurofeedback treatments in children with ADHD: an updated meta-analysis of randomized controlled trials. Front Hum Neurosci. 2014 Nov 13;8:906. doi: 10.3389/fnhum.2014.00906. eCollection 2014. PMID 25431555
- [Background] Heidbreder R. ADHD symptomatology is best conceptualized as a spectrum: a dimensional versus unitary approach to diagnosis. Atten Defic Hyperact Disord. 2015 Dec;7(4):249-69. doi: 10.1007/s12402-015-0171-4. Epub 2015 May 10. PMID 25957598
- [Result] Deiber MP, Hasler R, Colin J, Dayer A, Aubry JM, Baggio S, Perroud N, Ros T. Linking alpha oscillations, attention and inhibitory control in adult ADHD with EEG neurofeedback. Neuroimage Clin. 2020;25:102145. doi: 10.1016/j.nicl.2019.102145. Epub 2019 Dec 24. PMID 31911342